CLINICAL TRIAL: NCT00146367
Title: Evaluation of the Health Benefits of the Active Living Every Day Physical Activity Program Among Persons With Arthritis
Brief Title: Evaluation of the Active Living Every Day Exercise Program for People With Arthritis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of North Carolina (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCCDPHP-0444; CDC-NCCDPHP-MM-0444
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2005-09

CONDITIONS: Arthritis
Keywords: arthritis; osteoarthritis; rheumatoid arthritis; rheumatic disease; exercise; physical activity; physical function; disability
MeSH Terms: conditions — Arthritis; Osteoarthritis; Arthritis, Rheumatoid; Rheumatic Diseases; Motor Activity

INTERVENTIONS:
Behavioral: Active Living Every Day

SUMMARY:
The primary goal of this study is to assess the effectiveness and feasibility of the Active Living Every Day Physical Activity Program (ALED) for people with arthritis. This project is designed to evaluate the effectiveness of the ALED program in changing arthritis-related health outcomes and to investigate the feasibility of conducting the ALED program in a public health setting.

DETAILED DESCRIPTION:
Evidence has shown that regular moderate-intensity physical activity improves symptoms and function in persons with arthritis. A 20-week behavior-based program was developed by the Cooper Institute, Brown University, and Human Kinetics to help people with sedentary lifestyles become and stay physically active. A randomized trial evaluated the effectiveness and efficacy of a similar program on which Active Living Every Day is based (ALED) on cardiovascular disease risk factors, cost-effectiveness, and cardiorespiratory fitness. However, the current research supporting ALED is limited for people with arthritis. The primary goal of this study is to assess the effectiveness and feasibility of the Active Living Every Day Physical Activity Program (ALED) for people with arthritis. The primary goal will be accomplished through a twenty week randomized controlled trial conducted with 400 participants residing in the 17 Area Agencies on Aging housed in the Councils of Government in North Carolina, including both urban and rural counties. This project is designed to evaluate the effectiveness of the ALED program in changing arthritis-related health outcomes and to investigate the feasibility of conducting the ALED program in a public health setting.

Objectives:

1. To demonstrate that the ALED program can increase physical activity and fitness levels among people with arthritis.
2. To demonstrate that the Active Living Every Day has arthritis-specific benefits.
3. To evaluate the feasibility of disseminating the Active Living Every Day program through the NC public health network.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported arthritis or chronic joint symptoms
* Currently exercising less than 3 times per week
* Plan to be in community for at least 1 year
* Physician release for participation in physical activity

Exclusion Criteria:

* Pregnancy
* Non-English speaking
* Cognitive impairment
* Serious medical condition where exercise is contradindicated
* Severe physical or mental impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355
Dates: Start 2004-01; Study Completion 2005-10

PRIMARY OUTCOMES:
Physical Activity Level measured via CHAMPS instrument at baseline and 20 weeks
Physical Fitness Level measued via 2 minute step test at baseline and 20 weeks

SECONDARY OUTCOMES:
Functional status measured via HAQ at baseline and 20 weeks
Arthritis Self-efficacy measured at baseline and 20 weeks
Health-related Quality of Life measured at baseline, 20 weeks, 6 months and 12 months
Pain, fatigue and stiffness VAS at baseline and 20 weeks
Activities of Daily Living measured at baseline, 20 weeks, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Hootman, PhD, Study Chair — Centers for Disease Control and Prevention; Leigh F Callahan, PhD, Principal Investigator — University of North Carolina, Chapel Hill